CLINICAL TRIAL: NCT03860246
Title: Screening for Atrial Fibrillation in High-Risk Nursing Home Residents
Brief Title: Atrial Fibrillation Screening in Nursing Homes
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Anne Curtis, SUNY Distinguished Professor, State University of New York at Buffalo
Other Study IDs: STUDY00001737
Record Dates: First submitted 2019-02-14; First posted 2019-03-01 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Portable ECG monitor — Recording of ECG rhythm on a portable monitor (Kardia Mobile)

SUMMARY:
This study was designed to screen high risk patients in nursing homes for atrial fibrillation with intermittent electrocardiogram (ECG) recordings using a portable, smartphone-based, mobile ECG recording device (Kardia Mobile, AliveCor, Inc.). The investigators hypothesized that screening patients with 2 or more risk factors for atrial fibrillation would yield a higher incidence of atrial fibrillation compared to prior studies.

DETAILED DESCRIPTION:
This is a prospective study that enrolled 245 residents from 15 participating nursing homes with ≥2 risk factors for atrial fibrillation. All residents gave informed consent or had a legally appointed representative who could consent on their behalf. Exclusion criteria included residents with a prior diagnosis of atrial fibrillation, continuous rhythm monitoring over the past year, and pacemaker or implantable cardioverter defibrillator in situ.

Screening was performed using the smartphone-based, mobile ECG recording device. Thirty second rhythm recordings were obtained on each resident on four different occasions within a month. All tracings were reviewed by a cardiologist and, in the case of any uncertainty, the diagnosis of atrial fibrillation was confirmed by an electrophysiologist. When atrial fibrillation was detected in a resident (primary endpoint), no further rhythm recordings were performed and the resident's nursing facility was then notified of the diagnosis. Further evaluation and treatment were directed by the resident's primary care physician.

All data were stored on a secure encrypted server with password protection. The investigators used chi-square and t-test analyses to determine if there were significant differences in demographic variables or risk factors for atrial fibrillation between residents with and without atrial fibrillation. Logistic regression analysis determined if any combination of risk factors was predictive of a positive atrial fibrillation screen.

ELIGIBILITY:
Inclusion Criteria:

Nursing home residents with ≥2 of the following risk factors for atrial fibrillation:

* age ≥75 years
* female sex
* obstructive sleep apnea
* peripheral vascular disease
* diabetes mellitus
* obesity (body mass index [BMI] >30 kg/m2)
* hypertension
* congestive heart failure

Exclusion Criteria:

* prior diagnosis of AF
* continuous rhythm monitoring over the past year
* pacemaker or implantable cardioverter defibrillator in situ

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: nursing home residents
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
atrial fibrillation | 30 days
  number of participants with atrial fibrillation on any of four rhythm recordings

CONTACTS AND LOCATIONS:
Overall Officials: Anne B Curtis, MD, Principal Investigator — University at Buffalo
Locations (1):
- CTRC, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No